CLINICAL TRIAL: NCT04736784
Title: Effect of High Nitrate Vegetable Juice Supplementation on Plasma Nitrate and Blood Pressure in Healthy Adults: a Pilot Randomised Crossover Intervention in Healthy Volunteers
Brief Title: Effect of High Nitrate Vegetable Juice Supplementation on Plasma Nitrate and Blood Pressure in Healthy Adults
Acronym: NIVJUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Jayne Woodside, PhD, Professor, Queen's University, Belfast
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: QUB 16.60
Record Dates: First submitted 2021-01-21; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Blood Pressure
Keywords: nitrate rich juices; blood pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot juice (Experimental): 115 ml of beetroot juice per day for seven days
  Interventions: Other: Food-based - beetroot juice
- Leafy green vegetable juice (Experimental): 250 ml of green leafy vegetable juice per day for seven days
  Interventions: Other: Food-based - leafy green vegetable juice

INTERVENTIONS:
Other: Food-based - beetroot juice — Beetroot juice containing approximately 340 mg nitrate daily
  Arms: Beetroot juice
Other: Food-based - leafy green vegetable juice — Leafy green vegetable juice containing approximately 340 mg nitrate daily
  Arms: Leafy green vegetable juice

SUMMARY:
Aims: The aim of this study is to carry out a randomised crossover intervention study examining the effect of two different high nitrate vegetable juices on plasma nitrate levels and blood pressure (BP) in healthy adults.

Objectives: 1) to conduct a pilot cross-over randomized intervention study testing the hypothesis that the health benefits of two different high nitrate vegetable juices products will be similar; 2) to measure the volunteers' BP as the primary outcome; and 3) to collect biological samples over the course of this study for the measurement of proposed biomarkers of nutritional status, including plasma nitrate.

DETAILED DESCRIPTION:
In this study, it is hypothesized that oral supplementation with different vegetable juices (beetroot and green leafy vegetable) juice, with similar nitrate content, over a one week period, will decrease BP in healthy volunteers to a similar extent.

Plan of Investigation: This study will be a randomised, controlled, crossover (2 groups) trial of beetroot juice and green leafy vegetable juice.

Participants A total of 16 healthy volunteers will be recruited (male and female), according to the stated inclusion and exclusion criteria.

Recruitment Subjects will be screened and recruited from the general population through advertisement, through local community groups and staff intranet postings (university setting). The investigators have established mechanisms for recruiting from these populations that have proven to be effective in previous studies.

Study design Following screening, eligible participants will give informed written consent. Participants will be randomized, using computer-generated random numbers, to two groups.

Before starting the intervention (one week before), participants will be asked to complete a four day food diary.

Participants will consume one of the stated interventions daily (in the evening) for one week. Then, the participant will follow their normal diet and will not consume nitrate-rich juices for two weeks (washout period). In the fourth week, participants will consume the alternative intervention to that already consumed - beetroot juice or green leafy vegetables juice for a further one week.

Intervention products The beetroot juice will be Organic beetroot and apple juice (James White Drinks Ltd, UK), while the leafy green vegetable juice will be Leanandgreen (Cold Pressed Juice) composed of 30% celery, 30% cucumber, 15% romaine, 15% spinach, 5% kale, 2.5% ginger and 2.5% lemon (B. Fresh, UK). Both juices are available at Sainsbury's supermarket.

Both juices contain 5.5 mmol nitrate with different amount of the other nutrients. 250 ml of green leafy vegetable juice and 115 ml of beetroot juice will provide 5.5 mmol of nitrate daily to the participants.

Juices will provided to the volunteers by the researcher before the intervention week and both juices will have expiry dates that are beyond the intervention duration.

Other lifestyle practices Participants will be asked to not change any other part of their diet and to keep physical activity, alcohol, and caffeine and water source normal. Participants will be asked to avoid using mouthwash during the intervention weeks, as this can interfere with nitrate metabolism.

Justification for one-week intervention period. Inorganic nitrate and BP will respond quickly to the intervention, so a one week intervention period will be sufficiently long to ensure that participants will reach a steady state with regard to nitrate status.

Study assessments (for participant characterisation, in addition to primary and secondary outcome data collection as described) During each intervention week participants will be asked to complete a further four day food diary. Participants will also attend the Centre for Public Health (CPH) to give a blood sample and have BP measured at the start and end of each intervention period. Anthropometric data (weight and height) will also be obtained by standard procedures and BMI will be calculated as weight in kg divided by the squared height in metres.

Blood samples (20 ml) will be drawn from the antecubital vein and immediately separated and stored for the proposed assays detailed below. All blood samples will be stored at -70°C until analysis.

Power As this is a pilot study, power calculations have not been conducted.

Statistical analysis Statistical analysis will be carried out using SPSS for Windows, version 17. A medical statistician within CPH will give statistical advice where required. Analysis of this two-period crossover study will be carried out according to the Hills & Armitage method. If there are no significant period or carry-over effects, which will be tested for, paired samples t-tests will be used to compare the intervention group.

Data protection issues: Data collected in association with this study will be anonymised and archived in password-protected study databases. All biological samples collected will be anonymised.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Aged 30-65 years

Exclusion Criteria:

* Diabetes mellitus
* An acute coronary syndrome or transient ischaemic attack within the past 3 months
* Special dietary requirements, food sensitivities or vegetarian/ vegan diet by choice
* Oral anticoagulation therapy
* Recent beetroot juice (or other nitrate) supplementation.
* BMI>35 kg/m2
* Excessive alcohol consumption ( >14 U/week for men and women)
* Current smoker
* Pregnancy/ lactation
* Medical conditions or dietary restrictions that would substantially limit ability to complete the study requirements

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Blood pressure (clinic-based) | At baseline
  Clinic-based blood pressure using automated, calibrated blood pressure monitor, measured twice from the right arm, using an automated Omron sphygmomanometer, with the participant sitting quietly for at least five minutes.
Blood pressure (clinic-based) | After seven days
  Clinic-based blood pressure using automated, calibrated blood pressure monitor, measured twice from the right arm, using an automated Omron sphygmomanometer, with the participant sitting quietly for at least five minutes.
Blood pressure (home-assessed) | Pre juice consumption during the intervention
  An automated BP monitor (Omron M2Basic, Omron Healthcare) will be provided to each participant to measure daily resting BP at home. Participants will be asked to conduct duplicate measurements, in a seated position prior to juice consumption and at 2 hours after juice drinking and they will be trained on how to use the monitor, with an emphasis on the correct positioning of the cuff and arm. In addition, written instructions on measuring BP will be provided. Participants will be provided with a record sheet to record their measurements.
Blood pressure (home-assessed) | Two hours post juice consumption during the intervention
  An automated BP monitor (Omron M2Basic, Omron Healthcare) will be provided to each participant to measure daily resting BP at home. Participants will be asked to conduct duplicate measurements, in a seated position prior to juice consumption and at 2 hours after juice drinking and they will be trained on how to use the monitor, with an emphasis on the correct positioning of the cuff and arm. In addition, written instructions on measuring BP will be provided. Participants will be provided with a record sheet to record their measurements.

SECONDARY OUTCOMES:
Serum nitrate and nitrite concentrations | At baseline
  Serum concentrations of nitrate and nitrite. Total Nitric Oxide, nitrate and nitrite in plasma will be determined by an automated ELISA method (R&D Systems).
Serum nitrate and nitrite concentrations | After seven days
  Serum concentrations of nitrate and nitrite. Total Nitric Oxide, nitrate and nitrite in plasma will be determined by an automated ELISA method (R&D Systems).
Participant views on interventions | At end of the seven day intervention
  Acceptability and ease of consumption assessed via questionnaire with Likert scale responses

CONTACTS AND LOCATIONS:
Overall Officials: Jayne Woodside, Principal Investigator — Queen's University, Belfast
Locations (1):
- Centre for Public Health, Queen's University Belfast, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No